CLINICAL TRIAL: NCT04161417
Title: Precision-Panc Master Protocol: Personalising Treatment For Pancreatic Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Judith Dixon-Hughes (Other)
Collaborators: Cancer Research UK (Other); NHS Greater Glasgow and Clyde (Other)
Responsible Party: Sponsor-Investigator, Judith Dixon-Hughes, Project Manager, University of Glasgow
Organization: University of Glasgow (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: GN17on293
Record Dates: First submitted 2019-10-24; First posted 2019-11-13 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Neoplasms Pancreatic
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Intervention Model Description: The study is seen as interventional as patients may have more tissue taken at diagnositic biopsy than if they were not part of the trial or may have an extra biopsy if there is not enough material available from their diagnostic biopsy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Biopsy Material Required for Registration (Other): The Precision-Panc Master Protocol aims to recruit, consent and screen patients with pancreatic cancer
  Interventions: Other: Patients with suspected or confirmed pancreatic cancer will be be asked to provide biopsy material for molecular profiling

INTERVENTIONS:
Other: Patients with suspected or confirmed pancreatic cancer will be be asked to provide biopsy material for molecular profiling — Patients with suspected or confirmed pancreatic cancer will be be asked to provide biopsy material for molecular profiling. This will enable patient enrolment into a currently available PRIMUS study

SUMMARY:
The Precision-Panc Master Protocol is a "portal" protocol for patients with known or suspected pancreatic cancer to be accrued through multiple centres in the UK, with the option of being subsequently enrolled into PRIMUS (Pancreatic canceR Individualised Multi-arm Umbrella Studies) examining different treatment regimens and/or biomarker development. Eligible patients will undergo tumour biopsy and blood collection prospectively for molecular profiling at a central laboratory and the results may be used to inform enrolment to PRIMUS studies.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age >16 years).
* Either:

  * Presence of a hypodense pancreatic mass highly suspicious of primary pancreatic cancer with or without distant metastasis as assessed by a Pancreatic Multi-Disciplinary Team (MDT).

Or

o Histologically or cytologically confirmed pancreatic ductal adenocarcinoma and its variants.

* Patient is willing and able to undergo additional tumour biopsy (from the primary or a metastatic site) aimed at obtaining sufficient tissue for molecular profiling if this is required.
* Patient is deemed suitable to receive chemotherapy and/or radiotherapy, and/or surgery pending stage of disease at presentation.
* Patient is deemed potentially eligible for a currently open PRIMUS study
* Patient has signed informed consent for screening research tumour biopsy (Consent 1).
* Patient has signed informed consent for Precision-Panc Master Protocol molecular profiling (Consent 2).

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2500 (Estimated)
Dates: Start 2017-11-28 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Proving that patients with pancreatic cancer can have their tissue molecularly assessed and be followed up in a clinical trial setting | At end of study (5 years)
  The number of patients screened and registered to the master protocol will be recorded. The number of patients who we are able to molecular assess will be recorded and all patients will be followed up in the master protocol until death.

SECONDARY OUTCOMES:
Overall Survival | From date of registration until date of death from any cause, assessed up to 5 years
  To assess the overall survival (OS) in patients enrolled in Precision-Panc and relate this to molecular profile information.
Number of participants with biopsy related adverse events as assesed by CTCAE v4.03 | At time of biopsy, usually within one week of screening
  To assess the safety of obtaining tumour biopsies suitable for molecular profiling within a standard patient treatment pathway.

OTHER OUTCOMES:
Progression Free Survival | At time of progression (this is estimated at around 6-9 months for this group of patients)
  To assess the progression-free survival (PFS) in patients enrolled in Precision-Panc and relate this to molecular profile information

CONTACTS AND LOCATIONS:
Overall Officials: David Chang, Principal Investigator — University of Glasgow; Juan Valle, Principal Investigator — University of Manchester
Locations (33):
- United Kingdom (33):
  - Aberdeen Royal Infirmary, Aberdeen
  - Northern Ireland Cancer Centre, Belfast
  - Queen Elizabeth Hospital, Birmingham
  - Royal Bournemouth Hospital, Bournemouth
  - Bristol Oncology Centre, Bristol
  - Addenbrooke's Hospital, Cambridge
  - Castle Hill Hospital, Cottingham
  - Ninewells Hospital, Dundee
  - Western General, Edinburgh
  - Glasgow Royal Infirmary, Glasgow
  - Huddersfield Royal Infirmary, Huddersfield
  - Raigmore Hospital, Inverness
  - St James's Hospital, Leeds
  - Royal Liverpool Hospital, Liverpool
  - Guy's Hospital, London
  - Imperial College Healthcare Trust, London
  - King's College Hospital, London
  - Royal Free London Hospital, London
  - Royal Marsden Hospital, London
  - St Bart's Hospital, London
  - St George's Hospital, London
  - University College London Hospital, London
  - Manchester Royal Infirmary, Manchester
  - The Christie, Manchester, Manchester
  - Milton Keynes Hospital, Milton Keynes
  - Freeman Hospital, Newcastle
  - Nottingham Hospitals NHS Trust, Nottingham
  - Churchill Hospital, Oxford
  - Pool Hospital, Poole
  - Weston Park, Sheffield
  - University Hospital Southampton, Southampton
  - Morriston Hospital, Swansea
  - Royal Albert Edward Infirmary, Wigan

IPD SHARING:
Plan to Share IPD: Yes
When the clinical study report at end of study is complete all data will be available to other researchers. Researchers should contact study Trial Management Group for access. All genomic data will be made available through ICGC ARGO.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: On study completion
Access Criteria: Request to TMG

REFERENCES:
- [Derived] Saha A, Wadsley J, Sirohi B, Goody R, Anthony A, Perumal K, Ulahanan D, Collinson F. Can Concurrent Chemoradiotherapy Add Meaningful Benefit in Addition to Induction Chemotherapy in the Management of Borderline Resectable and Locally Advanced Pancreatic Cancer?: A Systematic Review. Pancreas. 2023 Jan 1;52(1):e7-e20. doi: 10.1097/MPA.0000000000002215. PMID 37378896